CLINICAL TRIAL: NCT00701766
Title: An Open, Randomised Clinical Phase I/IIa Trial to Investigate the Maximum Tolerated Dose, Efficacy, Safety and Pharmacokinetics of Repeated Three-week Courses of a Single Dose i.v. BI 2536 on Day 1 in Comparison to Single Doses i.v. BI 2536 on Days 1, 2 and 3 in Patients Over 60 Years of Age With Refractory or Relapsed Acute Myeloid Leukaemia
Brief Title: BI 2536 Infusional Treatment in Patients Over 60 Years of Age With Refractory or Relapsed Acute Myeloid Leukaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1216.20; EudraCT No:2006-000613-38
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2013-10

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BI 2536

INTERVENTIONS:
Drug: BI 2536

SUMMARY:
The present trial will be performed to determine the MTD and to evaluate the efficacy of BI 2536 in the treatment of elderly patients with relapsed or refractory AML. Different schedules will be compared to identify the better dosing schedule for the further development programme of BI 2536. Dose escalation starting with the maximum tolerated dose previously determined in patients with advanced solid cancers will be performed to determine the maximum tolerated dose for AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 60 years of age
* Patient with confirmed AML (except for APL) according to the WHO definition who relapsed after or are refractory to prior chemotherapy
* Leukocyte count <= 25,000 /mcl (25 x 10e9/Liter)
* Patient not eligible for intensive treatment options
* Life expectancy >= 2 months
* Eastern co-operative oncology group performance score of 2 or less
* Signed written informed consent consistent with international conference on harmonisation - good clinical practice (ICH-GCP) and local legislation

Exclusion Criteria:

* Patient with acute promyelocytic leukaemia (APL, AML of the French-American-British (FAB) classification subtype M3)
* Hypersensitivity to the trial drug or the excipients
* Secondary malignancy requiring therapy
* Known central nervous system involvement
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal, or AST or ALT greater than 5 times the upper limit of normal in case of known liver involvement
* Bilirubin greater than 1.5 mg/dl (> 26 mcmol/l, SI unit equivalent)
* Serum creatinine greater than 2.0 mg/dl
* Concomitant intercurrent illness, which would compromise the evaluation of efficacy or safety of the trial drug, e.g. active severe infection, unstable angina pectoris or cardiac arrhythmia
* Psychiatric illness or social situation that would limit compliance with trial requirements
* Concomitant therapy, which is considered relevant for the evaluation of the efficacy or safety of the trial drug
* Chemotherapy (except hydroxyurea) or immunotherapy or treatment with any other investigational drug within the past four weeks prior to treatment with the trial drug
* Persistence of toxicities of prior anti-leukaemia therapies which are deemed to be clinically relevant
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception during the trial (hormonal contraception, intrauterine device, condom with spermicide, etc.)
* Patient unable to comply with the protocol

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose Best objective response | 3 weeks, throughout the study period

SECONDARY OUTCOMES:
Event free survival, Overall survival, Remission duration, BI 2536 plasma concentrations, Incidence and intensity of adverse events graded according to CTCAE, PD, Incidence of DLT | throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (9):
- Austria (2):
  - 1216.20.43001 Boehringer Ingelheim Investigational Site, Innsbruck
  - 1216.20.43002 Boehringer Ingelheim Investigational Site, Vienna
- Germany (7):
  - 1216.20.49006 Boehringer Ingelheim Investigational Site, Bonn
  - 1216.20.49002 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1216.20.49003 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1216.20.49004 Boehringer Ingelheim Investigational Site, Hannover-Heideviertel
  - 1216.20.49007 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1216.20.49005 Boehringer Ingelheim Investigational Site, Münster
  - 1216.20.49001 Boehringer Ingelheim Investigational Site, Ulm